CLINICAL TRIAL: NCT00453492
Title: A Multicenter, Prospective, Randomized, 2-Way Crossover, Open-Label Study pn Postmenopausal Women With Osteoporosis Examining Subject Satisfaction and Compliance When Risedronate Sodium (Actonel) in Administered 35mg Once a Week or 5mg Once Daily
Brief Title: Risedronate Sodium in Post Menopausal Osteoporosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Procter and Gamble (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HMR4003B_4036
Record Dates: First submitted 2007-03-28; First posted 2007-03-29 (Estimated); Last update posted 2008-03-11 (Estimated); Status verified 2008-03

CONDITIONS: Osteoporosis, Postmenopausal
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Risedronic Acid

INTERVENTIONS:
Drug: risedronate sodium

SUMMARY:
The primary objective is to compare subject satisfaction of once a week dosing of 35 mg Actonel to once daily dosing of 5 mg Actonel in postmenopausal osteoporotic women.

The secondary objectives are to measure compliance (50 % drug taken), and persistence, [and urinary NTx (N-telopeptides) (optional)].

ELIGIBILITY:
Inclusion Criteria:

* Five years or greater postmenopausal who present with a diagnosis of postmenopausal osteoporosis based on standard clinical practice criteria.
* Subjects must discontinue bisphosphonates, calcitonin, fluoride, glucocorticoids (≥ 5 mg prednisone or equivalent per day) and hormone replacement therapy including estrogen-related compounds at least 6 months prior to randomization. During the study, these drugs are not permitted other than the study medication, Actonel.
* Other concomitant medications should be kept to a minimum, but if the drugs are considered necessary for the subject's welfare and are unlikely to interfere with study medication, they may be given at the discretion of the Investigator.

Exclusion criteria :

* Had a history of cancer within the past 5 years. Relatively benign skin malignancies, such as basal cell carcinoma or squamous cell carcinoma, are not an exclusion criteria if the subject has been in remission for at least 6 months prior to enrollment.
* Diagnosis of hypocalcemia, hyperparathyroidism, and hyperthyroidism.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 55 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246
Dates: Start 2004-01

PRIMARY OUTCOMES:
Measurement of subject satisfaction using a questionnaire at 12 and 24 weeks and a tablets counts at 12 and 24 weeks.
Optional: the effects of Actonel on bone resorption will be assessed by a change of urinary NTx, after 12 and 24 weeks of treatment as compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Edibe Taylan, Study Director — Sanofi-aventis, Turkey
Locations (1):
- Sanofi-Aventis, Istanbul, Turkey (Türkiye)